CLINICAL TRIAL: NCT03438916
Title: Hemodynamic Alterations in Liver Cirrhosis Validated by Non-invasive MRI Compared to Invasive Assessment: Can MRI and Echocardiography Predict the Pharmacological Response of Non-selective Beta-blocker in Patients With Cirrhosis?
Brief Title: MRI to Assess the Effect of Non-selective Beta-blocker in Patients With Cirrhosis
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Flemming Bendtsen, Professor, MD, Hvidovre University Hospital
Other Study IDs: 16048475
Record Dates: First submitted 2018-02-10; First posted 2018-02-20 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Portal Hypertension; Cirrhosis; Esophageal Varices; Gastric Varices Bleeding; Varice Bleed; Liver Diseases; Liver Cirrhosis
Keywords: Non-selective beta-blocker; Pharmacological respons; Magnetic Resonance Imaging; Hemodynamic assessments; Echocardiography; MR-elastography; Propranolol; Liver vein catheterization
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; Esophageal and Gastric Varices; Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard clinical blood tests and pertinent bioactive substances is measured in blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Standardization and new therapeutic treatments of variceal bleeding has significantly reduced the mortality the last 25 years, but there is still a high 6-week mortality around 15-20% and 1-year mortality of about 40%. Cirrhotic patients without prophylactic treatment suffer a risk of 60% of re-bleeding within the first year after the first bleeding episode. Variceal ligation and NSBB are the standard therapy as secondary prophylaxis, while only non-selective beta-blocker (NSBB) is offered as first-line therapy in primary prophylaxis. If portal pressure is reduced to a value below 12 mmHg or by 20% (10% if assessed by intravenous administrations), the risk of bleeding is substantially reduced, but not all patients respond to the treatment with propranolol (40-50%). Hence, patients who are non-responders to NSBB should be offered alternative treatment with e.g. carvedilol, which is a combined alpha-beta-receptor blocker or endoscopic band ligation. Currently, the response to NSBB is assessed invasively during a liver vein catheterization (LVC). Unfortunately, only a few centres in the world can perform this procedure and there are no reliable non-invasive alternatives to assess the respond to NSBB, which is of extreme importance, since non-responders have three fold increased risk of a new variceal bleeding episode.

Aim:

In general the aim of the project is to develop faster and non-invasive methods to evaluate portal hypertension and individual pharmacological response of NSBB in patients with cirrhosis. Furthermore, we expect to detect changes in liver and spleen stiffness as measured by MR-Elastography (MRE) after NSBB and that these depend on the drug-related effects on portal pressure.

Study design and patients:

39 patients with cirrhosis and esophageal varices that require NSBB (propranolol) treatment.

Patients are assessed with LVC, MR-scans, echocardiography and biochemical tests. LVC is the gold standard method to test if patients respond to propranolol treatment. At visit 1. the response to NSBB is defined as a reduction of HVPG ≥10%, or to a HVPG< 12mmHg after intravenous NSBB administrations during LVC. MRI-scan with intraveneus NSBB administration is performed at visit 2. Minimum 5 days of NSBB wash out between visit 1 and 2.

DETAILED DESCRIPTION:
MR-elastography and Phase Contrast MRI compared to LVC

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and esophageal varices that require NSBB treatment
* Patients of more than 18 and less than 78 years of age
* Patients with a portal pressure HVPG ≥ 12mmHg

Exclusion Criteria:

* Patients who are unable to give informed consent
* Patients with absolute contraindication for MRI
* Patients with absolute contraindication for NSBB
* Pregnant women
* Patient with severe hemodynamic comorbidity

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 39 patients with cirrhosis and esophageal varices that require NSBB (propranolol) treatment.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
NSBB response defined as a reduction in HVPG >10% or HVPG <12 mmHG after intraveneus NSBB administrations compared to flow (mL/min) in splanchnic vessels | after 20 minutes respons time
  To assess if changes in MR flow induced with NSBB (propranolol) administrations can predict the changes in HVPG after NSBB administration (NSBB respons) assessed by LVC

SECONDARY OUTCOMES:
MR-elastography | after 20 minutes
  To assess the liver and spleen stiffness (kPa) with MRE before and after intraveneus NSBB administration

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bendtsen, Professor, Principal Investigator — Professor
Locations (1):
- Centre of Gastroenterology, Dept. of medicine. Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Danielsen KV, Nabilou P, Wiese SS, Hove JD, Bendtsen F, Moller S. Effect of beta-blockers on multiple haemodynamics in cirrhosis: A cross-over study by MR-imaging and hepatic vein catheterization. Liver Int. 2023 Oct;43(10):2245-2255. doi: 10.1111/liv.15664. Epub 2023 Jun 30. PMID 37387503
- [Derived] Danielsen KV, Hove JD, Nabilou P, Yin M, Chen J, Zhao M, Kallemose T, Teisner AS, Siebner HR, Ehman RL, Moller S, Bendtsen F. Using MR elastography to assess portal hypertension and response to beta-blockers in patients with cirrhosis. Liver Int. 2021 Sep;41(9):2149-2158. doi: 10.1111/liv.14981. Epub 2021 Jun 16. PMID 34060714